CLINICAL TRIAL: NCT06712667
Title: The Effect of Coffee on People with High Intensity Exercise and the Characteristics of Caffeine Metabolism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, John R. Speakman, Professor, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SIAT IRB240915H0915
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: Coffee; Caffeine; Exercise; Caffeine metabolism
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Water (Placebo Comparator): The participants will drink 200 ml water.
  Interventions: Other: Caffeine content
- Decaffeinated coffee (Experimental): The participants will drink 200 ml decaffeinated coffee.
  Interventions: Other: Caffeine content
- Coffee (Experimental): The participants will drink 200 ml coffee, the caffeine content is 200 mg.
  Interventions: Other: Caffeine content

INTERVENTIONS:
Other: Caffeine content — Participants will drink the same volume of water or coffee with different amounts of caffeine.

SUMMARY:
The purpose of this project is to explore the relationship between the effect of coffee on exercise performance and caffeine metabolism.

DETAILED DESCRIPTION:
The investigators will study the relationship between the impact of coffee on exercise and caffeine metabolism. The investigators will recruit healthy elite athletes. Participants will be forbidden to consume stimulant drinks such as coffee for 24 hours before the experiment. When the participants arrive at the lab on the day of the experiment, they will sign an informed consent form, a health history questionnaire and a daily coffee consumption questionnaire. Each participant does six rides, with one day of caffeine washout before each ride. In all trials, each participant will ride at the same time of day. Before riding, drink 200 ml water, decaffeinated coffee or coffee in random order, and the caffeine content of coffee is 200 mg. After 60 minutes of drinking, they start riding, after the completion of the riding, the subjects perceived and judged the perception between the baseline load and the comparison load. After the completion of the judgment, the next level of stimulus parameters will randomly generated to conduct the experiment. Each person conducted 6 groups of intervention experiments. Changes in average exercise performance, heart rate, electrocardiogram and body temperature will be observed after drinking decaffeinated coffee or coffee compared with drinking water. The concentration of caffeine and its metabolites in urine before and after drinking within 3 hours will be measured by liquid chromatography-mass spectrometry (LC-MS) or gas chromatography-mass spectrometry (GC-MS).

ELIGIBILITY:
Inclusion Criteria:

Healthy adults 18-40 years old

Exclusion Criteria:

Diabetes Hypoglycemia Gout Osteoporosis Gastric ulcer Pancreatitis Intestinal obstruction Blood phobia Pathological hypo or hyper tension Impaired glucose tolerance Claustrophobia HIV,etc.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Exercise performance | On the experimental day, it lasts 2 weeks.
  After the completion of the riding, the subjects perceived and judged the perception between the baseline load and the comparison load.
Urine metabolites | On the experimental day, it lasts 2 weeks.
  The contents of metabolites will be measured by gas chromatography-mass spectrometry (GC-MS) and liquid chromatography-mass spectrometry (LC-MS ).

SECONDARY OUTCOMES:
Body temperature | On the experimental day, it lasts 2 weeks.
  Body temperature of participants will be measured by ear temperature gun.
Electrocardiogram (ECG) | On the experimental day, it lasts 2 weeks.
  ECG of participants will be measured by Amu ECG belt, the changes in P wave, PR interval, PR segment, QRS wave group, J point, ST segment, T wave, QT interval, and U wave will be observe.
Blood pressure | On the experimental day, it lasts 2 weeks.
  Systolic and diastolic blood pressure of participants will be measured by Omron digital sphygmomanometer.
Height | The morning of the first day of the experiment, 5 mins
  Height will be measured by seca 217 stable stadiometer. Subjects wearing no shoes.
Body weight | The morning of the first day of the experiment, 5 mins
  Fasting body weight will be measured by Bioimpedance Analysis (TANITA, MC-980).
Fat mass | The morning of the first day of the experiment, 10 mins
  Fat mass will be measured by Magnetic Resonance Imaging (Shanghai united imaging, uMR 790 ).
Fat free mass | The morning of the first day of the experiment, 10 mins
  Fat free mass will be measured by Bioimpedance Analysis (Tanita, MC-980).
Bone mass | The morning of the first day of the experiment, 10 mins
  Bone mass will be measured by Dual Energy X-ray Absorptiometry (Horizon Wi).
Heart rate | 2 weeks
  Heart rate will be measured by heart rate belt.
Waist circumferences | The morning of the first day of the experiment,10 mins
  Waist circumferences will be measured using a whole body laser scanner (TG2000-F).

CONTACTS AND LOCATIONS:
Overall Officials: John R Speakman, PhD, Study Chair — Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Locations (1):
- Shenzhen Institute of Advanced Technology, Chinese Academy of Sciences, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No